CLINICAL TRIAL: NCT00049361
Title: A Phase II Study Of Whole-Brain Radiation Therapy With Thalidomide And Temozolomide In Patients With Newly Diagnosed Brain Metastases
Brief Title: Radiation Therapy Plus Thalidomide and Temozolomide in Treating Patients With Newly Diagnosed Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: REBACDR0000258057; CCCWFU-91102; NCI-5883
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Brain and Central Nervous System Tumors; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: adult tumors metastatic to brain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Temozolomide; Thalidomide; Radiotherapy

INTERVENTIONS:
Drug: temozolomide
Drug: thalidomide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Combining whole-brain radiation therapy with thalidomide and temozolomide may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining whole-brain radiation therapy with thalidomide and temozolomide in treating patients who have newly diagnosed brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall median survival time of patients with newly diagnosed brain metastases treated with whole-brain radiotherapy in combination with thalidomide and temozolomide.
* Determine the radiographic response rate, median time to tumor progression, and median time to neurologic response and progression in patients treated with this regimen.
* Determine the cause of death of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Assess quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients undergo radiotherapy daily 5 days a week for 3 weeks. Beginning on the day before the first radiation treatment, patients receive oral thalidomide once daily and oral temozolomide once daily for 21 days. Patients continue to receive thalidomide daily for up to 2 years in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, 1 and 3 months after completing radiotherapy, and then every 3 months thereafter.

Patients are followed at 1 and 3 months and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 62 patients will be accrued for this study within 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed extracranial primary malignancy or brain metastases
* At least 1 brain metastasis with at least 1 unresected lesion that is measurable by contrast-enhanced MRI
* No evidence of spinal drop metastases or spread to noncontiguous meninges
* No lymphoma, small cell lung cancer, or germ cell tumor

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 4 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin less than 1.5 mg/dL
* SGPT and/or SGOT no greater than 2 times upper limit of normal

Renal

* Creatinine no greater than 1.5 mg/dL
* BUN no greater than 25 mg/dL

Other

* Able to be regularly followed
* No sensory neuropathy greater than grade 2
* No other major medical illnesses that would preclude study
* No neurologic or psychiatric impairments that would preclude study
* No active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use at least 1 highly effective and 1 additional effective method of contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No other concurrent chemotherapy during and for 4 weeks after study

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to head or neck
* No prior stereotactic radiosurgery
* Concurrent radiotherapy to extracranial sites of underlying malignancy allowed

Surgery

* Prior craniotomy allowed if completed within the past 10-28 days

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01-01 (Actual); Primary Completion 2004-12-07 (Actual); Study Completion 2004-12-07 (Actual)

PRIMARY OUTCOMES:
Overall median survival

SECONDARY OUTCOMES:
Radiographic response rate as assessed by MRI and RECIST one-dimensional criterion at 1 month, 3 months, and every 3 months thereafter
Median time to tumor progression
Median time to neurologic response and progression
Cause of death at median time
Quality of life as assessed by FACT-BT, FACT-F, and Beck Depression Inventory at 1 month, 3 months, and every 3 months thereafter
Toxicity as assessed by NCI Common Toxicity Criteria (CTC) version 2.0 for up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Volker W. Stieber, MD, Study Chair — Wake Forest University Health Sciences
Locations (5):
- United States (5):
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina